CLINICAL TRIAL: NCT02358031
Title: A Phase 3 Clinical Trial of Pembrolizumab (MK-3475) in First Line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Pembrolizumab (MK-3475) for First Line Treatment of Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck (MK-3475-048/KEYNOTE-048)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-048; MK-3475-048 (Other: MSD); KEYNOTE-048 (Other: MSD); 2014-003698-41 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2); chemotherapy, 5-fluorouracil, cisplatin, carboplatin
MeSH Terms: conditions — Head and Neck Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Carboplatin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab Monotherapy (Pembro Mono) (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years).
  Interventions: Biological: Pembrolizumab
- Pembrolizumab + Chemotherapy (Pembro Combo) (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years); plus cisplatin 100 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]); plus 5-FU 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-FU
- Cetuximab + Chemotherapy (Control) (Active Comparator): Participants receive cetuximab on Day 1 at a dose of 400 mg/m^2 IV, and then 250 mg/m^2 IV on Day 1 of each subsequent week until disease progression or unacceptable toxicity; plus cisplatin 100 mg/m^2 IV or carboplatin AUC 5 IV (Investigator's choice) on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months] for platinum-based therapy); plus 5-FU 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: 5-FU; Biological: Cetuximab

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years).
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Chemotherapy (Pembro Combo); Pembrolizumab Monotherapy (Pembro Mono)
Drug: Cisplatin — Cisplatin 100 mg/m^2 IV on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
  Arms: Cetuximab + Chemotherapy (Control); Pembrolizumab + Chemotherapy (Pembro Combo)
Drug: Carboplatin — Carboplatin at a target AUC 5 IV on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
  Arms: Cetuximab + Chemotherapy (Control); Pembrolizumab + Chemotherapy (Pembro Combo)
Drug: 5-FU — 5-FU 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
  Arms: Cetuximab + Chemotherapy (Control); Pembrolizumab + Chemotherapy (Pembro Combo)
Biological: Cetuximab — Cetuximab on Day 1 at a dose of 400 mg/m^2 IV, and then 250 mg/m^2 IV on Day 1 of each subsequent week until disease progression or unacceptable toxicity
  Arms: Cetuximab + Chemotherapy (Control)

SUMMARY:
Participants with recurrent or metastatic (R/M) squamous cell cancer of the head and neck (HNSCC) will be randomly assigned to receive pembrolizumab monotherapy [pembro mono], pembrolizumab plus chemotherapy with a platinum-based drug (cisplatin or carboplatin) and 5-Fluorouracil (5-FU) [pembro combo], or cetuximab plus a platinum-based drug (cisplatin or carboplatin) and 5-FU [control]. The overall primary study hypotheses are as follows in all participants and in participants with Programmed Cell Death Ligand 1 (PD-L1) positive expression defined by Combined Positive Score (CPS) ≥1 and CPS ≥20: 1) pembrolizumab monotherapy prolongs progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) assessed by Blinded Independent Central Review (BICR) and prolongs overall survival (OS) compared to standard treatment, and 2) pembrolizumab combination with chemotherapy prolongs PFS per RECIST 1.1 assessed by BICR and prolongs OS compared to standard treatment.

DETAILED DESCRIPTION:
The 12 primary superiority hypotheses will be evaluated by comparing the pembro mono arm or pembro combo arm separately to the control arm, for PFS and OS in all first line (1L) R/M HNSCC participants and in 1L R/M HNSCC participants with positive PD-L1 expression (PD-L1 CPS ≥1 and CPS ≥20).

Per protocol, response/progression or adverse events (AEs) that occur during the second pembrolizumab course will not be counted towards efficacy outcome measures or safety outcome measures, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed recurrent or metastatic head and neck squamous cell carcinoma considered incurable by local therapies
* No prior systemic therapy administered in the recurrent or metastatic setting (with the exception of systemic therapy completed > 6 months prior if given as part of multimodal treatment for locally advanced disease)
* Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx. Participants may not have a primary tumor site of nasopharynx (any histology)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Can provide tissue for PD-L1 biomarker analysis from a core or excisional biopsy (fine needle aspirate is not sufficient): A newly obtained biopsy (within 90 days prior to start of study treatment) is preferred but an archival sample is acceptable.
* Have results from testing of human papillomavirus (HPV) status for oropharyngeal cancer
* Female participants of childbearing potential should have a negative pregnancy test and must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication
* Male participants must agree to use an adequate method of contraception starting with the first dose of study medication through 180 days after the last dose of study medication

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent
* Has progressive disease (PD) within six (6) months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC
* Radiation therapy (or other non-systemic therapy) within 2 weeks prior to randomization or not fully recovered from adverse events due to a previously administered treatment
* Currently participating and receiving study therapy, or participated in a study of an investigational agent and received study therapy, or used an investigational device within 4 weeks of the first dose of study medication
* Life expectancy of <3 months and/or has rapidly progressing disease
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication (physiologic doses of corticosteroids may be approved after consultation with the Sponsor)
* Diagnosed and/or treated additional malignancy within 5 years prior to randomization with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers
* Has had an allogeneic tissue/solid organ transplant
* Active central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of study medication
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or previously participated in Merck MK-3475 clinical trial
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Received a live vaccine within 30 days of planned start of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Tahara M, Greil R, Rischin D, Harrington KJ, Burtness B, de Castro G, Psyrri A, Brana I, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Ishak WZW, Lin J, Gumuscu B, Lerman N, Soulieres D. Pembrolizumab with or without chemotherapy in recurrent or metastatic head and neck squamous cell carcinoma: 5-year follow-up from the randomized phase III KEYNOTE-048 study. Eur J Cancer. 2025 May 15;221:115395. doi: 10.1016/j.ejca.2025.115395. Epub 2025 Apr 4. PMID 40262400
- [Derived] Oridate N, Takahashi S, Tanaka K, Shimizu Y, Fujimoto Y, Matsumoto K, Yokota T, Yamazaki T, Takahashi M, Ueda T, Hanai N, Yamaguchi H, Hara H, Yoshizaki T, Yasumatsu R, Nakayama M, Shiga K, Fujii T, Mitsugi K, Takahashi K, Nohata N, Gumuscu B, Lerman N, Tahara M. First-line pembrolizumab with or without chemotherapy for recurrent or metastatic head and neck squamous cell carcinoma: 5-year follow-up of the Japanese population of KEYNOTE-048. Int J Clin Oncol. 2024 Dec;29(12):1825-1839. doi: 10.1007/s10147-024-02632-x. Epub 2024 Oct 9. PMID 39382718
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] Takahashi S, Oridate N, Tanaka K, Shimizu Y, Fujimoto Y, Matsumoto K, Yokota T, Yamazaki T, Takahashi M, Ueda T, Hanai N, Yamaguchi H, Hara H, Yoshizaki T, Yasumatsu R, Nakayama M, Shiga K, Fujii T, Mitsugi K, Takahashi K, Nohata N, Gumuscu B, Swaby RF, Tahara M. First-line pembrolizumab +/- chemotherapy for recurrent/metastatic head and neck cancer: Japanese subgroup of KEYNOTE-048. Int J Clin Oncol. 2022 Dec;27(12):1805-1817. doi: 10.1007/s10147-022-02233-6. Epub 2022 Oct 20. PMID 36264378
- [Derived] Harrington KJ, Burtness B, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Lin J, Gumuscu B, Swaby RF, Rischin D. Pembrolizumab With or Without Chemotherapy in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: Updated Results of the Phase III KEYNOTE-048 Study. J Clin Oncol. 2023 Feb 1;41(4):790-802. doi: 10.1200/JCO.21.02508. Epub 2022 Oct 11. PMID 36219809
- [Derived] Rischin D, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Ishak WZW, Hong RL, Mendoza RG, Jia L, Chirovsky D, Norquist J, Jin F, Burtness B. Pembrolizumab alone or with chemotherapy for recurrent or metastatic head and neck squamous cell carcinoma: Health-related quality-of-life results from KEYNOTE-048. Oral Oncol. 2022 May;128:105815. doi: 10.1016/j.oraloncology.2022.105815. Epub 2022 Apr 2. PMID 35381576
- [Derived] Burtness B, Rischin D, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Ge J, Swaby RF, Gumuscu B, Harrington K. Pembrolizumab Alone or With Chemotherapy for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma in KEYNOTE-048: Subgroup Analysis by Programmed Death Ligand-1 Combined Positive Score. J Clin Oncol. 2022 Jul 20;40(21):2321-2332. doi: 10.1200/JCO.21.02198. Epub 2022 Mar 25. PMID 35333599
- [Derived] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26083&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with first line recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) were recruited to examine the efficacy and safety of pembrolizumab monotherapy (pembro mono) versus pembrolizumab plus chemotherapy (pembro combo) versus cetuximab plus chemotherapy (control).
Pre-assignment Details: Of 1228 participants screened, 882 were randomized to the pembro mono arm, pembro combo arm, or control arm. 22 participants in the control arm that enrolled during an enrollment pause of the pembro combo arm were excluded from efficacy comparisons between the pembro combo arm and control arm.
  Per protocol, response/progression or adverse events (AEs) that occurred during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab Monotherapy (Pembro Mono): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years). Qualified participants who received the first course of pembrolizumab but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule of 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
- Pembrolizumab + Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years); plus cisplatin 100 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]); plus 5-Fluorouracil (5-FU) 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]). Qualified participants who received the first course of pembrolizumab but continued to experience disease progression may have, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule of 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
- Cetuximab + Chemotherapy (Control): Participants received cetuximab on Day 1 at a dose of 400 mg/m^2 IV, and then 250 mg/m^2 IV on Day 1 of each subsequent week until disease progression or unacceptable toxicity; plus cisplatin 100 mg/m^2 IV or carboplatin AUC 5 IV (Investigator's choice) on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months] for platinum-based therapy); plus 5-FU 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
Period: Overall Study
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Started | 301 | 281 | 300
Treated | 300 | 276 | 287
Pembro Mono v Control Efficacy Analyses | 301 | 0 | 300
Pembro Combo v Control Efficacy Analyses | 0 | 281 | 278
Received Second Course of Pembrolizumab | 8 | 6 | 0
Completed | 2 | 1 | 0
Not Completed | 299 | 280 | 300
Not completed — Death | 253 | 237 | 266
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 19 | 14 | 18
Not completed — Sponsor Decision | 26 | 28 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control) | Total
Number analyzed (Participants) | 301 | 281 | 300 | 882
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (9.4) | 60.7 (9.8) | 61.0 (10.0) | 61.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 57 | 39 | 147
  Male | 250 | 224 | 261 | 735
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 45 | 44 | 135
  Not Hispanic or Latino | 233 | 213 | 231 | 677
  Unknown or Not Reported | 22 | 23 | 25 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 6 | 14
  Asian | 58 | 60 | 54 | 172
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 11 | 6 | 21
  White | 219 | 203 | 224 | 646
  More than one race | 12 | 4 | 9 | 25
  Unknown or Not Reported | 3 | 0 | 1 | 4
Eastern Cooperative Group (ECOG) Performance Status [Count of Participants; unit: Participants] — An ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) was required for inclusion in the trial.
  Participants
    ECOG = 0 | 118 | 110 | 117 | 345
    ECOG = 1 | 183 | 171 | 183 | 537
Human Papillomavirus (HPV) Status [Count of Participants; unit: Participants] — HPV status for oropharynx cancer as determined by p16 immunohistochemistry (IHC) (positive vs. negative); HPV status for participants without oropharynx cancer was considered HPV negative.
  Participants
    HPV Positive | 63 | 60 | 67 | 190
    HPV Negative | 238 | 221 | 233 | 692
PD-L1 TPS Status [Count of Participants; unit: Participants] — The Programmed Cell Death Ligand 1 (PD-L1) Tumor Proportion Score (TPS) Status indicates the degree by which participants tumors stain positive for PD-L1 by IHC staining (i.e. strongly positive or not strongly positive). Participants with a TPS ≥50% were classified as PD-L1 "strongly positive" and participants with a TPS <50% were classified as "not strongly positive."
  Participants
    Strongly Positive | 67 | 66 | 66 | 199
    Not Strongly Positive | 234 | 215 | 234 | 683
PD-L1 CPS ≥1 Status [Count of Participants; unit: Participants] — The PD-L1 Combined Positive Score (CPS) Status indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by IHC. The number of participants with CPS<1 and CPS≥1 at baseline is presented. Participants with a CPS<1 were classified as PD-L1 negative and participants with a CPS≥1 were classified as PD-L1 positive.
  Participants
    CPS<1 | 44 | 39 | 45 | 128
    CPS ≥1 | 257 | 242 | 255 | 754
PD-L1 CPS ≥20 Status [Count of Participants; unit: Participants] — The PD-L1 CPS Status indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by IHC. The number of participants with CPS<20 and CPS ≥20 at baseline is presented.
  Participants
    CPS <20 | 167 | 154 | 175 | 496
    CPS ≥20 | 133 | 126 | 122 | 381
    Missing | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pembro Combo vs Control: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the Intent-To-Treat (ITT) population. PFS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm. Per protocol, PFS was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: All participants in the ITT population randomized to either the pembro combo arm or control arm during active enrollment were analyzed. 22 participants in the control arm enrolled during an enrollment pause of the pembro combo arm were excluded. Per protocol, pembro mono arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab Monotherapy (Pembro Mono): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years).
- Pembrolizumab + Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years); plus cisplatin 100 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]); plus 5-Fluorouracil (5-FU) 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 281 | 278
Months |  | 4.9 [4.7 to 6.1] | 5.2 [4.9 to 6.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); PFS in all participants of the pembro combo arm was compared to PFS in all participants of the control arm to address the sixth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.21211, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.78 to 1.11]

2. Primary Outcome: Pembro Combo vs Control: PFS Per RECIST 1.1 by BICR in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the ITT population. PFS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm with PD-L1 biomarker positive expression defined by immunohistochemistry (IHC) as Combined Positive Score ≥1 (hereafter referred to as CPS ≥1). Per protocol, PFS was compared separately between CPS ≥1 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: Participants in the ITT population randomized to either pembro combo arm or control arm during active enrollment with CPS ≥1 were analyzed. 20 participants in control arm enrolled during an enrollment pause of the pembro combo arm were excluded. Per protocol, pembro mono arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 242 | 235
Months |  | 5.1 [4.7 to 6.2] | 5.0 [4.8 to 6.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); PFS in CPS ≥1 participants of the pembro combo arm was compared to PFS in CPS ≥1 participants of the control arm to address the fifth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.03697, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.02]

3. Primary Outcome: Pembro Combo vs Control: PFS Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the ITT population. PFS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm with PD-L1 biomarker positive expression defined by IHC as Combined Positive Score ≥20 (hereafter referred to as CPS ≥20). Per protocol, PFS was compared separately between CPS ≥20 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: Participants in the ITT population randomized to either pembro combo arm or control arm during active enrollment with CPS ≥20 were analyzed. 12 participants in control arm enrolled during an enrollment pause of the pembro combo arm were excluded. Per protocol, pembro mono arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 126 | 110
Months |  | 5.8 [4.7 to 7.6] | 5.3 [4.9 to 6.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); PFS in CPS ≥20 participants of the pembro combo arm was compared to PFS in CPS ≥20 participants of the control arm to address the fourth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG and HPV status; Test type: Superiority; p = 0.02951, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG and HPV status; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.58 to 1.01]

4. Primary Outcome: Pembro Combo vs Control: Overall Survival (OS) in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm. Per protocol, OS was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 281 | 278
Months |  | 13.0 [10.9 to 14.7] | 10.7 [9.3 to 11.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); OS in all participants of the pembro combo arm was compared to OS in all participants of the control arm to address the fourteenth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.00025, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.60 to 0.87]

5. Primary Outcome: Pembro Combo vs Control: OS in Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥1. Per protocol, OS was compared separately between CPS ≥1 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 242 | 235
Months |  | 13.6 [10.7 to 15.5] | 10.4 [9.1 to 11.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); OS in CPS ≥1 participants of the pembro combo arm was compared to OS in CPS ≥1 participants of the control arm to address the twelfth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.00002, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.53 to 0.80]

6. Primary Outcome: Pembro Combo vs Control: OS in Participants With PD-L1 CPS ≥20
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro combo arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥20. Per protocol, OS was compared separately between CPS ≥20 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 126 | 110
Months |  | 14.7 [10.3 to 19.3] | 11.0 [9.2 to 13.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); OS in CPS ≥20 participants of the pembro combo arm was compared to OS in CPS ≥20 participants of the control arm to address the eleventh primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG and HPV status; Test type: Superiority; p = 0.00044, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG and HPV status; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.45 to 0.82]

7. Primary Outcome: Pembro Mono vs Control: PFS Per RECIST 1.1 by BICR in All Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. PFS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm. Per protocol, PFS was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: All participants in the ITT population randomized to either the pembro mono arm or control arm during active enrollment were analyzed. Per protocol, pembro combo arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 301 | 0 | 300
Months | 2.3 [2.2 to 3.3] |  | 5.2 [4.9 to 6.1]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); PFS in all participants of the pembro mono arm was compared to PFS in all participants of the control arm to address the third primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.99830, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [1.09 to 1.53]

8. Primary Outcome: Pembro Mono vs Control: PFS Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. PFS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥1. Per protocol, PFS was compared separately between CPS ≥1 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: All participants in the ITT population randomized to either the pembro mono arm or control arm during active enrollment with CPS ≥1 were analyzed. Per protocol, pembro combo arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 257 | 0 | 255
Months | 3.2 [2.2 to 3.4] |  | 5.0 [4.8 to 6.0]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); PFS in CPS ≥1 participants of the pembro mono arm was compared to PFS in CPS ≥1 participants of the control arm to address the second primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.89580, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.94 to 1.36]

9. Primary Outcome: Pembro Mono vs Control: PFS Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. PFS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥20. Per protocol, PFS was compared separately between CPS ≥20 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: All participants in the ITT population randomized to either the pembro mono arm or control arm during active enrollment with CPS ≥20 were analyzed. Per protocol, pembro combo arm was compared to control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 133 | 0 | 122
Months | 3.4 [3.2 to 3.8] |  | 5.3 [4.8 to 6.3]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); PFS in CPS ≥20 participants of the pembro mono arm was compared to PFS in CPS ≥20 participants of the control arm to address the first primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG and HPV status; Test type: Superiority; p = 0.46791, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG and HPV status; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.76 to 1.29]

10. Primary Outcome: Pembro Mono vs Control: OS in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm. Per protocol, OS was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 301 | 0 | 300
Months | 11.5 [10.3 to 13.4] |  | 10.7 [9.3 to 11.7]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); OS in all participants of the pembro mono arm was compared to OS in all participants of the control arm to address the tenth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.01985, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.99]

11. Primary Outcome: Pembro Mono vs Control: OS in Participants With PD-L1 CPS ≥1
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥1. Per protocol, OS was compared separately between CPS ≥1 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 257 | 0 | 255
Months | 12.3 [10.8 to 14.3] |  | 10.3 [9.0 to 11.5]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); OS in CPS ≥1 participants of the pembro mono arm was compared to OS in CPS ≥1 participants of the control arm to address the eighth primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, HPV status and PD-L1 status; Test type: Superiority; p = 0.00133, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG, HPV status and PD-L1 status; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.61 to 0.90]

12. Primary Outcome: Pembro Mono vs Control: OS in Participants With PD-L1 CPS ≥20
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro mono arm was compared to the control arm as a pre-specified primary analysis of the ITT population. OS is reported here for the first course of treatment, for all participants in the pembro mono arm and control arm with PD-L1 biomarker positive expression defined by IHC as CPS ≥20. Per protocol, OS was compared separately between CPS ≥20 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 133 | 0 | 122
Months | 14.8 [11.5 to 20.6] |  | 10.7 [8.8 to 12.8]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); OS in CPS ≥20 participants of the pembro mono arm was compared to OS in CPS ≥20 participants of the control arm to address the seventh primary hypothesis. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG and HPV status; Test type: Superiority; p = 0.00010, Regression, Cox — One-sided p-value based on log-rank test stratified by ECOG and HPV status; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.44 to 0.78]

13. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among All Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 281 | 278
Percentage of Participants |  | 44.7 [38.8 to 50.5] | 44.9 [38.9 to 50.8]

14. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between CPS ≥1 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 242 | 235
Percentage of Participants |  | 44.9 [38.5 to 51.1] | 43.3 [36.9 to 49.6]

15. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between CPS ≥20 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 126 | 110
Percentage of Participants |  | 49.4 [40.3 to 57.9] | 47.2 [37.5 to 56.2]

16. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among All Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 281 | 278
Percentage of Participants |  | 17.2 [13.0 to 21.9] | 13.6 [9.8 to 18.1]

17. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between CPS ≥1 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 242 | 235
Percentage of Participants |  | 19.7 [14.8 to 25.0] | 12.5 [8.6 to 17.3]

18. Secondary Outcome: Pembro Combo vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro combo arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between CPS ≥20 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 126 | 110
Percentage of Participants |  | 23.9 [16.7 to 31.7] | 14.0 [8.2 to 21.3]

19. Secondary Outcome: Pembro Combo vs Control: Objective Response Rate (ORR) Per RECIST 1.1 by BICR in All Participants
Description: ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants in the pembro combo arm and control arm. Per protocol, ORR was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 281 | 278
Percentage of Participants |  | 35.6 [30.0 to 41.5] | 36.3 [30.7 to 42.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); ORR in all participants of the pembro combo arm was compared to ORR in all participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.5740, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = -0.8, 95% CI 2-sided [-8.7 to 7.2]

20. Secondary Outcome: Pembro Combo vs Control: ORR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro combo arm and control arm. Per protocol, ORR was compared separately between CPS ≥1 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 242 | 235
Percentage of Participants |  | 36.4 [30.3 to 42.8] | 35.7 [29.6 to 42.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); ORR in CPS ≥1 participants of the pembro combo arm was compared to ORR in CPS ≥1 participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.4586, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = 0.5, 95% CI 2-sided [-8.2 to 9.1]

21. Secondary Outcome: Pembro Combo vs Control: ORR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥20
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro combo arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro combo arm and control arm. Per protocol, ORR was compared separately between CPS ≥20 participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 126 | 110
Percentage of Participants |  | 42.9 [34.1 to 52.0] | 38.2 [29.1 to 47.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); ORR in CPS ≥20 participants of the pembro combo arm was compared to ORR in CPS ≥20 participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1) and HPV status (Positive vs. Negative); Test type: Other; p = 0.2161, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = 5.0, 95% CI 2-sided [-7.5 to 17.4]

22. Secondary Outcome: Pembro Combo vs Control: Change From Baseline to Week 15 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100; a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 15 in the GHS/QoL combined score, for the first course of treatment, was compared between all participants of the pembro combo arm and the control arm as a pre-specified secondary analysis. Per protocol, change from baseline to Week 15 in the GHS/QoL combined score was compared separately between all participants of the pembro mono arm and control arm and is presented later in the record.
Time Frame: Baseline, Week 15
Population: Participants in pembro combo arm and control arm who received ≥1 dose of study drug and with EORTC-QLQ-C30 assessments available at baseline or post-baseline up to Week 15. 20 in control arm enrolled during enrollment pause of the pembro combo arm were excluded. Per protocol, pembro mono arm compared to control arm separately and not included here.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 268 | 259
Score on a Scale |  | 1.17 [-1.79 to 4.12] | 0.77 [-2.22 to 3.76]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); Change from baseline to Week 15 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro combo arm and the control arm. Comparison based on constrained longitudinal data analysis (cLDA) model with GHS/QoL score as response variable and treatment by visit interaction, stratification factors (ECOG [0 vs. 1], HPV status [Positive vs. Negative] and PD-L1 TPS status [Strongly Positive, Not Strongly Positive]) as covariates; Test type: Other; p = 0.839, constrained Longitudinal Data Analysis — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = 0.40, 95% CI 2-sided [-3.46 to 4.26]

23. Secondary Outcome: Pembro Combo vs Control: Time to Deterioration (TTD) in the EORTC QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Combined Score (Kaplan-Meier Method)
Description: EORTC-QLQ-C30 is a 30-item questionnaire to assess the QoL of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicating a better overall outcome. TTD in GHS/QoL defined as the time from baseline to the first onset of a ≥10 point decrease from baseline in GHS/QoL combined score, with confirmation. Per protocol, TTD in GHS/QoL combined score, for first course of treatment, was compared between all participants of pembro combo arm and control arm as a pre-specified secondary analysis; and TTD in GHS/QoL combined score was compared separately between all participants of pembro mono arm and control arm and is presented later in the record.
Time Frame: Baseline up to approximately 12 months
Population: All participants in the pembro combo arm and the control arm who completed the EORTC QLQ-C30 and had received ≥1 dose of study drug. 20 in the control arm enrolled during an enrollment pause of the pembro combo arm were excluded. Per protocol, the pembro mono arm was compared to the control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 270 | 260
Months |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); TTD in GHS/QoL combined score was compared between all participants of the pembro combo arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.9497, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.94 to 2.00]

24. Secondary Outcome: Pembro Combo vs Control: TTD in the EORTC QLQ- Head and Neck Module 35 (H&N35) Pain Score (Kaplan-Meier Method)
Description: EORTC QLQ-H&N35 is a 35-item questionnaire to assess QoL of head and neck cancer participants and consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. Participant responses to the Pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. TTD in EORTC QLQ-H&N35 Pain Score defined as the time from baseline to the first onset of a ≥10 point decrease from baseline, with confirmation. Per protocol, TTD in EORTC QLQ-H&N35 Pain Score, for the first course of treatment, was compared between all participants of pembro combo arm and control arm as a pre-specified secondary analysis. Also per protocol, TTD in EORTC QLQ-H&N35 Pain Score was compared separately between all participants of pembro mono arm and control arm and is presented later in the record.
Time Frame: Baseline up to approximately 12 months
Population: All participants in the pembro combo arm and control arm who completed the EORTC QLQ-H&N35 and had received ≥1 dose of study drug. 20 in the control arm enrolled during an enrollment pause of the pembro combo arm were excluded. Per protocol, the pembro mono arm was compared to the control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 268 | 260
Months |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); TTD in EORTC QLQ-H&N35 Pain Score was compared between all participants of the pembro combo arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.9476, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.93 to 2.02]

25. Secondary Outcome: Pembro Combo vs Control: TTD in the EORTC QLQ- H&N35 Swallowing Score (Kaplan-Meier Method)
Description: EORTC QLQ-H&N35 is a 35-item questionnaire developed to assess QoL of head and neck cancer participants and consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. Participant responses to the Swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicating more problems. TTD in EORTC QLQ-H&N35 Swallowing Score defined as the time from baseline to the first onset of a ≥10 point decrease from baseline, with confirmation. Per protocol, TTD in EORTC QLQ-H&N35 Swallowing Score, for the first course of treatment, was compared between all participants of pembro combo arm and control arm as a pre-specified secondary analysis; and compared separately between all participants of pembro mono arm and control arm and is presented later in the record.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 0 | 268 | 260
Months |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy (Pembro Combo) vs Cetuximab + Chemotherapy (Control); TTD in EORTC QLQ-H&N35 Swallowing Score was compared between all participants of the pembro combo arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.5836, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.69 to 1.59]

26. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among All Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 6
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 301 | 0 | 300
Percentage of Participants | 26.2 [21.4 to 31.3] |  | 45.7 [39.9 to 51.3]

27. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between CPS ≥1 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 6
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 257 | 0 | 255
Percentage of Participants | 28.7 [23.3 to 34.4] |  | 43.9 [37.6 to 49.9]

28. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 6 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 6 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 6 months was compared separately between CPS ≥20 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 6
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 133 | 0 | 122
Percentage of Participants | 33.0 [25.2 to 41.0] |  | 46.6 [37.5 to 55.2]

29. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among All Participants
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 301 | 0 | 300
Percentage of Participants | 17.6 [13.5 to 22.1] |  | 15.0 [11.2 to 19.4]

30. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥1
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between CPS ≥1 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 257 | 0 | 255
Percentage of Participants | 20.6 [15.9 to 25.8] |  | 13.6 [9.6 to 18.2]

31. Secondary Outcome: Pembro Mono vs Control: Percentage of Participants With PFS at 12 Months Per RECIST 1.1 by BICR Among Participants With PD-L1 CPS ≥20
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants with PFS (PFS rate) at 12 months is reported here, for the first course of treatment, out of all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro mono arm and control arm. Per protocol, the percentage of participants with PFS at 12 months was compared separately between CPS ≥20 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Month 12
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 133 | 0 | 122
Percentage of Participants | 23.5 [16.6 to 31.1] |  | 15.1 [9.3 to 22.2]

32. Secondary Outcome: Pembro Mono vs Control: ORR Per RECIST 1.1 by BICR in All Participants
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants in the pembro mono arm and control arm. Per protocol, ORR was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 301 | 0 | 300
Percentage of Participants | 16.9 [12.9 to 21.7] |  | 36.0 [30.6 to 41.7]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); ORR in all participants of the pembro mono arm was compared to ORR in all participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive , Not Strongly Positive); Test type: Other; p = 1.0000, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = -19.0, 95% CI 2-sided [-25.8 to -12.1]

33. Secondary Outcome: Pembro Mono vs Control: ORR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥1 in the pembro mono arm and control arm. Per protocol, ORR was compared separately between CPS ≥1 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 257 | 0 | 255
Percentage of Participants | 19.1 [14.5 to 24.4] |  | 34.9 [29.1 to 41.1]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); ORR in CPS ≥1 participants of the pembro mono arm was compared to ORR in CPS ≥1 participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 1.0000, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = -15.9, 95% CI 2-sided [-23.4 to -8.3]

34. Secondary Outcome: Pembro Mono vs Control: ORR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥20
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro mono arm was compared to the control arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR, for the first course of treatment, for all participants with PD-L1 biomarker positive expression defined by IHC as CPS ≥20 in the pembro mono arm and control arm. Per protocol, ORR was compared separately between CPS ≥20 participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Up to approximately 47 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 133 | 0 | 122
Percentage of Participants | 23.3 [16.4 to 31.4] |  | 36.1 [27.6 to 45.3]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); ORR in CPS ≥20 participants of the pembro mono arm was compared to ORR in CPS ≥20 participants of the control arm. The comparison was based on Miettinen & Nurminen method stratified by ECOG (0 vs. 1) and HPV status (Positive vs. Negative); Test type: Other; p = 0.9869, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = -12.8, 95% CI 2-sided [-23.8 to -1.5]

35. Secondary Outcome: Pembro Mono vs Control: Change From Baseline to Week 15 in the EORTC QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 15 in the GHS/QoL combined score, for the first course of treatment, was compared between all participants of the pembro mono arm and the control arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 15 in the GHS/QoL combined score was compared separately between all participants of the pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Baseline, Week 15
Population: All participants in the pembro mono arm and the control arm who received ≥1 dose of study drug and had EORTC-QLQ-C30 assessments available at baseline or post-baseline up to Week 15. Per protocol, the pembro combo arm was compared to the control arm separately and not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 294 | 0 | 279
Score on a Scale | 0.85 [-1.90 to 3.59] |  | 0.60 [-2.19 to 3.40]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); Change from baseline to Week 15 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro mono arm and the control arm. Comparison based on cLDA model with GHS/QoL score as response variable and treatment by visit interaction, stratification factors (ECOG [0 vs. 1], HPV status [Positive vs. Negative] and PD-L1 TPS status [Strongly Positive, Not Strongly Positive]) as covariates; Test type: Other; p = 0.893, constrained Longitudinal Data Analysis — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = 0.24, 95% CI 2-sided [-3.34 to 3.82]

36. Secondary Outcome: Pembro Mono vs Control: TTD in the EORTC QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: EORTC-QLQ-C30 is a 30-item questionnaire to assess the QoL of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicating a better overall outcome. TTD in GHS/QoL defined as the time from baseline to the first onset of a ≥10 point decrease from baseline in GHS/QoL combined score, with confirmation. Per protocol, TTD in GHS/QoL combined score, for the first course of treatment, was compared between all participants of pembro mono arm and control arm as a pre-specified secondary analysis; and compared separately between all participants of pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Baseline up to approximately 12 months
Population: All participants in the pembro mono arm and the control arm who completed the EORTC QLQ-C30 and had received ≥1 dose of study drug. Per protocol, the pembro combo arm was compared to the control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 294 | 0 | 280
Months | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); TTD in GHS/QoL combined score was compared between all participants of the pembro mono arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.9530, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.95 to 2.00]

37. Secondary Outcome: Pembro Mono vs Control: TTD in the EORTC QLQ- H&N35 Pain Score
Description: EORTC QLQ-H&N35 is a 35-item questionnaire developed to assess QoL of head and neck cancer participants and consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. Participant responses to the Pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicating more problems. TTD in EORTC QLQ-H&N35 Pain Score defined as the time from baseline to the first onset of a ≥10 point decrease from baseline, with confirmation. Per protocol, TTD in EORTC QLQ-H&N35 Pain Score, for the first course of treatment, was compared between all participants of pembro mono arm and control arm as a pre-specified secondary analysis. Also per protocol, TTD in EORTC QLQ-H&N35 Pain Score was compared separately between all participants of pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Baseline up to approximately 12 months
Population: All participants in the pembro mono arm and control arm who completed the EORTC QLQ-H&N35 and had received ≥1 dose of study drug. Per protocol, the pembro combo arm was compared to the control arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 295 | 0 | 280
Months | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); TTD in EORTC QLQ-H&N35 Pain Score was compared between all participants of the pembro mono arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.1501, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.53 to 1.21]

38. Secondary Outcome: Pembro Mono vs Control: TTD in the EORTC QLQ- H&N35 Swallowing Score
Description: EORTC QLQ-H&N35 is a 35-item questionnaire developed to assess QoL of head and neck cancer participants and consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. Participant responses to the Swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100; a higher score indicating more problems. TTD in EORTC QLQ-H&N35 Swallowing Score defined as the time from baseline to the first onset of a ≥10 point decrease from baseline, with confirmation. Per protocol, TTD in EORTC QLQ-H&N35 Swallowing Score, for the first course of treatment, was compared between all participants of pembro mono arm and control arm as a pre-specified secondary analysis; and compared separately between all participants of pembro combo arm and control arm and is presented earlier in the record.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 37
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 295 | 0 | 280
Months | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event. |  | NA [NA to NA] — NA=Median and 95% confidence interval limits not reached due to an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Cetuximab + Chemotherapy (Control); TTD in EORTC QLQ-H&N35 Swallowing Score was compared between all participants of the pembro mono arm and the control arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG (0 vs. 1), HPV status (Positive vs. Negative) and PD-L1 TPS status (Strongly Positive, Not Strongly Positive); Test type: Other; p = 0.8751, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.85 to 1.88]

39. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE, for the first course of treatment, was reported for each arm.
Time Frame: Up to approximately 47 months
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 300 | 276 | 287
Participants | 290 | 271 | 286

40. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that discontinued study drug due to an AE, for the first course of treatment, was reported for each arm.
Time Frame: Up to approximately 47 months
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + Chemotherapy (Pembro Combo) | Cetuximab + Chemotherapy (Control)
Number analyzed (Participants) | 300 | 276 | 287
Participants | 36 | 90 | 79

ADVERSE EVENTS:
Time Frame: Up to approximately 98 months
Description: All-Cause Mortality (ACM): all randomized participants. AEs: all randomized participants who got ≥1 dose of study drug. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs. Per protocol, ACM and AEs were collected and reported separately for pembrolizumab second course.
Groups:
- Pembrolizumab Monotherapy (First Course): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years).
- Pembrolizumab + Chemotherapy (First Course): Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 35 cycles (up to ~2 years); plus cisplatin 100 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum [up to ~4 months]); plus 5-FU 1000 mg/m^2/day IV continuous from Day 1-4 of each 3-week cycle (6 cycle maximum [up to ~4 months]).
- Pembrolizumab Monotherapy (Second Course): Qualified participants who received the first course of pembrolizumab monotherapy but continued to experience disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
- Pembrolizumab + Chemotherapy (Second Course): Qualified participants who received the first course of pembrolizumab in combination with chemotherapy but continued to experience disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
Arm/Group | Pembrolizumab Monotherapy (First Course) | Pembrolizumab + Chemotherapy (First Course) | Cetuximab + Chemotherapy (Control) | Pembrolizumab Monotherapy (Second Course) | Pembrolizumab + Chemotherapy (Second Course)
All-Cause Mortality (participants affected / at risk) | 260/301 | 242/281 | 282/300 | 5/8 | 5/6
Serious Adverse Events (participants affected / at risk) | 123/300 | 165/276 | 142/287 | 1/8 | 2/6
Other Adverse Events (participants affected / at risk) | 265/300 | 266/276 | 278/287 | 6/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (First Course) (N=300) | Pembrolizumab + Chemotherapy (First Course) (N=276) | Cetuximab + Chemotherapy (Control) (N=287) | Pembrolizumab Monotherapy (Second Course) (N=8) | Pembrolizumab + Chemotherapy (Second Course) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 14 (17) | 9 (11) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 17 (17) | 15 (16) | 0 (0) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 4 (6) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 8 (9) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Autoinflammatory disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Type III immune complex mediated reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Medical device site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 20 (25) | 23 (25) | 20 (24) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 5 (5) | 8 (10) | 3 (3) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (7) | 4 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 6 (7) | 5 (5) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery perforation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 1 (2) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurogenic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (First Course) (N=300) | Pembrolizumab + Chemotherapy (First Course) (N=276) | Cetuximab + Chemotherapy (Control) (N=287) | Pembrolizumab Monotherapy (Second Course) (N=8) | Pembrolizumab + Chemotherapy (Second Course) (N=6)
Anaemia (Blood and lymphatic system disorders) | 61 (82) | 153 (210) | 128 (251) | 2 (6) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 37 (57) | 41 (87) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 7 (10) | 9 (20) | 16 (58) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (14) | 90 (135) | 93 (194) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 74 (111) | 71 (148) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 17 (17) | 19 (21) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 55 (57) | 45 (48) | 18 (22) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 7 (7) | 5 (5) | 6 (10) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 9 (11) | 19 (27) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 11 (13) | 19 (24) | 1 (1) | 0 (0)
Apical granuloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 59 (62) | 101 (145) | 95 (134) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 44 (54) | 77 (121) | 96 (191) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 17 (18) | 20 (23) | 10 (12) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 15 (18) | 24 (28) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 20 (21) | 31 (37) | 27 (28) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 49 (58) | 140 (271) | 146 (273) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 7 (7) | 18 (18) | 14 (14) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 67 (104) | 77 (121) | 0 (0) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 33 (43) | 90 (155) | 77 (123) | 0 (0) | 0 (0)
Asthenia (General disorders) | 16 (16) | 46 (75) | 43 (64) | 0 (0) | 0 (0)
Fatigue (General disorders) | 81 (94) | 95 (133) | 101 (162) | 1 (1) | 1 (1)
Malaise (General disorders) | 6 (6) | 21 (25) | 8 (10) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 12 (15) | 80 (131) | 80 (137) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 12 (12) | 17 (18) | 18 (21) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 36 (41) | 41 (69) | 37 (46) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (6) | 7 (8) | 6 (8) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 4 (4) | 22 (24) | 17 (25) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 39 (55) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15) | 19 (22) | 12 (12) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 4 (5) | 3 (4) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (3) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 11 (12) | 14 (18) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (18) | 19 (23) | 22 (48) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 17 (22) | 20 (25) | 25 (37) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 12 (19) | 37 (61) | 24 (50) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 7 (16) | 2 (3) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 4 (4) | 6 (6) | 7 (10) | 2 (2) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 2 (4) | 3 (3) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 10 (16) | 15 (33) | 13 (34) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 50 (85) | 55 (106) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 53 (98) | 49 (80) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 42 (43) | 43 (50) | 59 (65) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 4 (6) | 36 (76) | 46 (110) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 44 (51) | 78 (101) | 81 (112) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 12 (12) | 16 (20) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 12 (12) | 17 (23) | 8 (9) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (28) | 15 (23) | 23 (42) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (10) | 17 (25) | 18 (49) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (9) | 6 (9) | 3 (14) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (11) | 23 (31) | 15 (22) | 1 (4) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 17 (23) | 22 (49) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (28) | 30 (43) | 53 (90) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (12) | 42 (62) | 115 (270) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 26 (31) | 34 (53) | 36 (72) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (10) | 12 (18) | 26 (45) | 0 (0) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (29) | 22 (32) | 18 (20) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 12 (15) | 12 (13) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 18 (22) | 28 (30) | 21 (26) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 14 (16) | 28 (34) | 39 (62) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 9 (9) | 18 (19) | 16 (19) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 36 (42) | 32 (39) | 24 (36) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 16 (18) | 8 (10) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 16 (17) | 7 (9) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 6 (7) | 3 (5) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 15 (15) | 12 (13) | 15 (18) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 21 (23) | 28 (31) | 24 (30) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (48) | 53 (65) | 37 (53) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 (43) | 19 (20) | 18 (27) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (11) | 22 (34) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (14) | 8 (10) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (15) | 21 (24) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 11 (11) | 6 (6) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 7 (8) | 4 (4) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 15 (15) | 15 (15) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 (9) | 1 (1) | 84 (130) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (16) | 10 (11) | 38 (49) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6) | 22 (37) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (39) | 24 (26) | 32 (51) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 31 (43) | 30 (37) | 112 (160) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (10) | 16 (24) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 38 (50) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 13 (14) | 18 (27) | 16 (19) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 6 (8) | 10 (11) | 21 (33) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02358031/Prot_SAP_001.pdf